CLINICAL TRIAL: NCT03234075
Title: Promoting Access to Renal Transplantation: Impact of a Patient-centered Regional Organization
Brief Title: Evaluation of a New Regional Organization to Promote Access to Renal Transplantation
Acronym: TRACE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL17_0022
Record Dates: First submitted 2017-07-26; First posted 2017-07-31 (Actual); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Renal Failure
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control group: Patients supported without regional organization for promotion of renal transplantation Setting : French Auvergne Rhone Alpes region and French Center region
- Intervention group: Patients supported with the regional organization for promotion of renal transplantation Setting : French Auvergne Rhone Alpes region
  Interventions: Other: Regional organization for promotion of renal transplantation

INTERVENTIONS:
Other: Regional organization for promotion of renal transplantation — Early identification of candidates for renal transplantation
  * with the help of a care coordinator Inform all patients appropriately about the techniques of renal function supplementation
  * delivered by expert patients and a care coordinator Assist the nephrologists in patient graft pathway
  * Multidisciplinary assessment of patients in dedicated web-conferencing meetings bringing together nephrologists and transplant team (" WebRCP of kidney transplant orientation")
  * Helping to carry out the pre-graft assessments of patients by a care coordinator
  Groups: Intervention group

SUMMARY:
Patients with terminal chronic kidney disease (CRD) need renal function supplementation, namely dialysis or renal transplantation. Transplantation is the most efficient and cost-effective treatment. Early and equitable access to transplantation is a public health issue. Access to transplantation is facilitated by early and systematic information and assessment of patients for inclusion in the national waiting list for transplantation prior to the onset of dialysis, and by the development of transplantation from living donors. In France, there are wide disparities in access to national waiting list registration and transplantation. One of the causes of these inequalities in access would be the disparity in referral practices to a transplant medical and surgical team authorized to register the individual on the national waiting list.

The aim of the TRACE study is to evaluate the impact of a new regional organization promoting renal transplantation on access to renal transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Patient older than 18 years and younger than 85 years.
* Entered in the French Network Epidemiology and Information in Nephrology register
* Renal function supplementation begun in 2013 -- 2014 (period before regional organization implementation) or in 2018 -- 2019 (period after regional organization implementation).

Exclusion Criteria:

- Patient followed in a Center of nephrology-dialysis or of Renal transplantation located outside French Auvergne Rhône Alpes or Center Regions.

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population participating in the study is composed of patients with a terminal Chronic Kidney Disease (CRD) requiring renal function supplementation.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidence rate of access to renal transplantation for patients with end-stage renal failure | At 24 months after initiation of renal function supplementation
  Access to renal transplantation is defined by:
  * Pre-emptive renal transplantation with living donor or deceased donor
  * Registration on the national waiting list for renal transplantation

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Transplantation, Groupement Hospitalier Edouard Herriot, Hospices Civils de Lyon, Lyon, France

IPD SHARING:
Plan to Share IPD: No